CLINICAL TRIAL: NCT03634995
Title: A Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunologic Effects of BMS-986256, and a Relative Bioavailability Study in Healthy Participants
Brief Title: An Investigational Study to Evaluate the Effects of Experimental Medication BMS-986256 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM026-002; 2017-003729-13 (EudraCT Number)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Dose (Experimental): Ascending single doses of BMS-986256
  Interventions: Drug: BMS-986256; Other: Placebo
- Multiple Dose (Experimental): Ascending multiple doses of BMS-986256
  Interventions: Drug: BMS-986256; Other: Placebo
- Sequential Dose (Experimental): Sequential multiple doses of BMS-986256
  Interventions: Drug: BMS-986256; Other: Placebo

INTERVENTIONS:
Drug: BMS-986256 — Specified dose on specified days
Other: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the effects of the experimental medication BMS-986256 in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Weight ≥ 50 kg and body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive at screening
* Participants must not be current users (within 6 months before screening) of tobacco or tobacco- or nicotine-containing products; they must also be willing to refrain from using any of these products during their participation in the study
* A negative QuantiFERON®-TB Gold test result at screening or documentation of a negative result within 3 months before screening

Exclusion Criteria:

* Previous participation in the current study or previous exposure within 6 weeks before study drug administration for non-biologics and 12 weeks before study drug administration for biologics
* Inability to tolerate oral medication
* Inability to tolerate venipuncture, or inadequate venous access

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Events (SAE) | Up to 46 days
Number of deaths | Up to 46 days
Number of clinically significant changes in ECG, vital signs, physical examination findings, or clinical laboratory assessments | Up to 44 days
Number of Adverse Events (AEs) leading to early discontinuation | Up to 44 days
Maximum concentration (Cmax) | Up to 44 days
Time of maximum concentration (Tmax) | Up to 44 days
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration [AUC(0-T)] | Up to 44 days
Area under the plasma concentration-time curve extrapolated to infinity [AUC(INF)] | Up to 44 days

SECONDARY OUTCOMES:
Terminal elimination rate constant (kel) | Up to 44 days
Terminal elimination half-life (T-half) | Up to 44 days
Apparent oral clearance (CL/F) | Up to 44 days
Metabolite ratio for AUC(INF) [MR(AUC[INF])] | Up to 44 days
Metabolite ratio of Cmax [MR(Cmax)] | Up to 44 days
Apparent volume of distribution at terminal phase (Vz/F) | Up to 44 days
Plasma concentration immediately prior to dosing (Ctrough) | Up to 44 days
Area under the plasma concentration-time curve over the dosing interval [AUC(TAU)] | Up to 44 days
Accumulation ratio of Ctrough [AR(Ctrough)] | Up to 44 days
Accumulation ratio of AUC(TAU) [AR(AUC[TAU])] | Up to 44 days
Accumulation ratio of Cmax [AR(Cmax)] | Up to 44 days
Metabolite ratio for AUC(TAU) [MR(AUC[TAU])] | Up to 44 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, Anaheim, California
  - PRA Health Science KK, Lenexa, Kansas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm